CLINICAL TRIAL: NCT05961423
Title: Robotic Versus Laparoscopic D3-D4 Lymphadenectomy for Patients With Advanced Colorectal Cancer… A Randomized Prospective Clinical Trial for the Comparison of Oncologic and Functional Outcomes
Brief Title: Robotic vs Laparoscopic D3-D4 Lymphadenectomy for Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Division of colorectal surgery, department of surgery, National Taiwan University Hospital, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202002011RINB
Record Dates: First submitted 2023-07-09; First posted 2023-07-27 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer
Keywords: Lymphadenectomy; Colorectal cancer; D3-D4
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Control group: laparoscopic surgery Interventional group: robotic surgery
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic surgery (No Intervention): The patients will undergoing laparoscopic surgery for the treatment of locally advanced colorectal cancer
- Robotic group (Active Comparator): The patients will undergoing robotic surgery for the treatment of locally advanced colorectal cancer
  Interventions: Procedure: Robotic surgery

INTERVENTIONS:
Procedure: Robotic surgery — The patient group undergoing robotic surgery for the treatment of locally advanced colorectal cancer
  Arms: Robotic group

SUMMARY:
Approximately one third of patients with colorectal cancer are diagnosed as locally advanced stage with metastasis to N3 - N4 lymph nodes requiring a D3 - D4 lymphadenectomy. Our previous study has indicated that, by laparoscopic approach, the extended abdomino-iliac lymphadenectomy, the so-called D3-D4 lymph node dissection, could be performed with quick convalescence and similar oncologic efficacy for the treatment of advanced recto-sigmoid cancer with metastatic lesions over N3-N4 lymph nodes, as compared with traditional open surgery. In the present study, the investigators will further compare the oncologic and functional outcomes of robotic versus laparoscopic approach in performing such challenging surgical procedures for patients with advanced colorectal cancer requiring a D3-D4 lymphadenectomy through a randomized prospective clinical trial.

DETAILED DESCRIPTION:
Approximately one third of patients with colorectal cancer are diagnosed as locally advanced stage with metastasis to N3 - N4 lymph nodes requiring a D3 - D4 lymphadenectomy. Our previous study has indicated that, by laparoscopic approach, the extended abdomino-iliac lymphadenectomy, the so-called D3-D4 lymph node dissection, could be performed with quick convalescence and similar oncologic efficacy for the treatment of advanced recto-sigmoid cancer with metastatic lesions over N3-N4 lymph nodes, as compared with traditional open surgery. In the present study, the investigators will further compare the oncologic and functional outcomes of robotic versus laparoscopic approach in performing such challenging surgical procedures for patients with advanced colorectal cancer requiring a D3-D4 lymphadenectomy through a randomized prospective clinical trial.

In the upcoming three years (2020/4/1-2023/3/31),consecutive recto-sigmoid cancer patients with metastasis to para- aortic lymph node will be screened and randomized to patient groups undergoing either robotic or laparoscopic D3-D4 lymph node dissection. The extent of D4 lymph node dissection includes extirpation of the extra-mesenteric lymphatic basin along bilateral common iliac arteries and veins, inferior vena cava, and abdominal aorta upward to the level just below the duodenal third portion and left renal vein, besides the traditional mesenteric dissection of paracolic (N1) lymph nodes, intermediate (N2) mesenteric lymph nodes, and lymph nodes around the root of inferior mesenteric artery (N3). The harvested lymph nodes were mapped and managed according to the Japanese guidelines. The metrics of surgical outcomes included: the number of harvested lymph nodes; time to recurrence of cancer after surgery; the length of operation time; blood loss; intra-operative and post-operative complications; and wound size. Functional recovery was evaluated by length of post-operative flatus passage, the restoration of urinary function, hospitalization, and degree of post-operative pain. A subjective-response standardized questionnaire was given to patients to assess disability, which included the number of days until return to partial activity, full activity, and work.

Since the current randomized prospective study in this field is still lack of, the investigators believe that this study will be of academic importance. And, clinically, the presented study can to help set up the standard operation procedures for such patient, and provide the level one evidence for National Health Insurance Administration in evaluating the reimbursement of HTA (high technology assessment) procedures.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proved adenocarcinoma located at upper rectum (above pelvic peritoneal reflection), recto-sigmoid junction, or distal sigmoid colon (generally 10 to 25 cm above anal verge). Only recto-sigmoid cancers above the peritoneal reflection were investigated because the lymphatic drainage of upper rectum and distal sigmoid colon was along the inferior mesenteric artery to the para-aortic area, and therefore the extent of surgical resection and lymph node mapping were standardized.
* Clinically TNM stage III cancers.
* Curative robotic or laparoscopic surgery.
* American Society of Anesthesiology (ASA) class I to III patients.
* Age between 50 and 75 years. This was because patients >50 years old are generally deemed to be over the reproductive age, and the D3 dissection was considered too aggressive for patients older than 75 years.
* Patients who are willing to receive minimally invasive surgical procedures to treat their rectosigmoid cancer.

Exclusion Criteria:

* Tumors located at other anatomic positions;
* Emergency or palliative surgery;
* Evidence of disseminated disease or adjacent organ invasion;
* Primary tumor mass ≥8 cm in diameter;
* Morbidly obese patients (body mass index ≥40 kg/m2);
* Previous major surgery of lower abdomen.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
The time to recurrence of cancer after curative resection | Up to 3 years
  The duration between the time of curative resection and the time to cancer recurrence

SECONDARY OUTCOMES:
the number of dissected lymph nodes | An average of 7 days
  The total numbers of lymph node harvested during the operation
The distribution of dissected lymph nodes | An average of 7 days
  The total numbers of lymph node harvested in different lymph node area during the operation
Functional recovery | Up to 6 months
  Functional questionnaire regarding fecal continence and bowel function will be completed by an assistant not aware of the randomization status of the patient right after completion of the manometric studies. Continence was recorded as Grade 1 (perfect continence), Grade 2 (incontinence of flatus), Grade 3 (occasional minor soiling), Grade 4 (frequent major soiling), and Grade 5 (total incontinence).
The overall costs of both minimally invasive surgical approaches | Through patients' discharge from hospital, an average of 7 days
  The total medical costs including medication fee and equipment fee are recorded.
Assessment of disability | 12 months
  The time for the patients after the operation to resume partial activity, full activity, and return to work will be recorded to evaluate the disability.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tung LIANG, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- Jin-Tung LIANG, Taipei, Taiwan